CLINICAL TRIAL: NCT03274089
Title: A Randomized Controlled Trial to Evaluate the Health Outcomes of Patients With Stable Chronic Disease Managed With a Healthcare Kiosk
Brief Title: Health Outcomes of Patients With Stable Chronic Disease Managed With a Healthcare Kiosk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Principal Investigator, Grace Ng Beng Hua, Family Physician, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1629027001
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Hypertension; Hyperlipidemia; Mixed; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Hyperlipoproteinemia Type II; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kiosk intervention group (Experimental)
  Interventions: Device: Kiosk intervention group
- Nurse clinician control group (No Intervention)

INTERVENTIONS:
Device: Kiosk intervention group — SEEK automates the management of patients with stable well-controlled chronic disease. SEEK has the following capabilities:
  * Collects patient information using patient-specific identification
  * Prompts the user for answers to screening questions for acute conditions
  * Measures relevant physiological parameters: blood pressure, height, weight; and calculates body mass index
  * Triages patients based on responses to screening questions, physiological parameters and blood test results
  * Provides recommendations to the patient on the care plan, self management and lifestyle choices
  Other Names: SEEK® MyHealthKiosk
  Arms: Kiosk intervention group

SUMMARY:
The chronic disease burden is increasing worldwide leading to a rise in the demand for primary healthcare and a shortage of primary care physicians. Addressing this shortage entails a multi-prong approach with innovations in care delivery, greater use of healthcare technology, and more efficient use of all healthcare providers on the care team.

We previously developed an interactive self-service healthcare kiosk (Self-empowering and enabling kiosk - SEEK® MyHealthKiosk) for the management of patients with stable chronic disease in the primary care setting. A feasibility study using SEEK showed high levels of acceptance and satisfaction from patients and healthcare providers.

The aim of this follow-up study is to evaluate the health outcomes of patients with stable chronic disease who are on kiosk management compared to patients who are on routine management by nurse clinicians. We hypothesize that patients who are managed by the kiosk continue to maintain good disease control that are comparable to patients who are managed by a nurse clinician.

DETAILED DESCRIPTION:
Patients who seek primary healthcare vary in their time and resource requirements. Patients with acute medical conditions or poorly controlled chronic disease typically require more time and attention compared to patients with stable chronic disease.

Patients with chronic disease routinely make follow-up visits to their primary care provider for assessment of their chronic disease status and for changes to their medications as necessary. Patients with well-controlled stable chronic disease may go through several visits to their primary care provider in 3 or 4-monthly intervals with little or no change to their medication regimen. These patients have to wait in line with the rest of the patient crowd for a doctor's consultation before getting their regular supply of medications. We hence saw the potential of replacing some of these physician visits with an automated healthcare kiosk so that if the disease condition of such patients remained stable, they can continue on their current medications without having to see a doctor.

We previously described the feasibility of using an automated healthcare kiosk (SEEK® MyHealthKiosk) for the management of patients with stable chronic disease in the primary care setting. We propose a follow-up study to show equivalence of health outcomes for patients managed with SEEK compared to the current standard of care. The study will be a 2-armed randomized controlled trial of 120 patients with stable chronic disease on 4-monthly follow-up visits over a 12-month period. Patients will be assigned randomly to intervention or control groups to receive kiosk or nurse management respectively. The main primary outcome measure is the overall chronic disease control of the patients. Other primary outcome measures are the blood pressure and low-density lipoprotein cholesterol levels for patients without diabetes; and blood pressure, low-density lipoprotein cholesterol and hemoglobin A1c levels for patients with diabetes. Secondary outcome measures are visit duration, patient satisfaction with the management process, health-related quality of life, and the occurrence of any adverse event.

The potential benefits from the use of SEEK are:

1. Appropriate stratification of patient care needs so that more time and resources can be channeled to patients with complex or acute needs;
2. Patient empowerment in the management of their chronic health conditions, with flexibility of self-care and monitoring and decreased dependency on healthcare providers;
3. Substitution of nurse clinicians for the management of stable chronic disease;
4. Reduction in the number of doctor visits per year for patients with stable chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* are between the ages of 21 and 75 years
* have at least one chronic medical condition that includes hypertension, hyperlipidemia, diabetes mellitus
* have blood pressure, low-density lipoprotein cholesterol (LDL-C) and HbA1c levels within the recommended targets according to the Ministry of Health Singapore clinical practice guidelines for their current and last follow-up visits
* are able to provide informed consent.

Exclusion Criteria:

* have serum creatinine more than 140 mmol/L (from tests done within the past year)
* have serum potassium less than 3.5 mmol/L or more than 5 mmol/L (from tests done within the past year)
* have overt proteinuria (urine protein:creatinine ratio more than 0.5)
* were discharged from hospital or specialist follow-up within the last 6 months
* have any pending laboratory or investigation result
* are scheduled for any laboratory investigation within the next 4 months (except HbA1c or panel test)
* have any new complaint related to their chronic medical conditions
* have a known history of white coat hypertension

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Disease control | 12 months
Blood pressure | 12 months
Low-density lipoprotein cholesterol | 12 months
Hemoglobin A1c | 12 months

SECONDARY OUTCOMES:
Visit duration | 8 months
Patient satisfaction questionnaire | 12 months
  The following areas of patient satisfaction will be scored on a Likert scale: convenience of visit schedule, location of kiosk or nurse consultation, appropriateness of management, duration of time spent in kiosk usage or nurse consultation, and the replacement of a doctor's visit by the kiosk or nurse clinician. Qualitative feedback will be captured via free-text inputs.
Adverse events | 12 months
Health-related quality of life questionnaire | 12 months
  Health-related quality of life will be assessed using the EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- SingHealth Polyclinics - Punggol, Singapore, Singapore

REFERENCES:
- [Derived] Ng G, Tan SW, Tan NC. Health outcomes of patients with chronic disease managed with a healthcare kiosk in primary care: protocol for a pilot randomised controlled trial. BMJ Open. 2018 Mar 23;8(3):e020265. doi: 10.1136/bmjopen-2017-020265. PMID 29574445